CLINICAL TRIAL: NCT00003120
Title: Phase III Randomized Trial of 12 Months vs. 3 Months of Paclitaxel in Patients With Advanced Ovarian Cancer Who Attain a Clinically Defined Complete Response (CR) Following Platinum/Paclitaxel-Based Chemotherapy
Brief Title: S9701 Paclitaxel in Treating Patients With Advanced Ovarian, Fallopian Tube, or Primary Peritoneal Cancer in Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065875; SWOG-S9701 (Other: SWOG); GOG-178 (Other: GOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paclitaxel 3 cycles (Active Comparator): paclitaxel given for 3 cycles
  Interventions: Drug: paclitaxel
- paclitaxel for 12 cycles (Experimental): paclitaxel given for 12 cycles
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel — 135 mg/m2 IV every 28 days
  Other Names: taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known whether giving paclitaxel for a shorter period of time is as effective as a standard course of treatment for advanced ovarian cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel given for 3 months with that of paclitaxel given for 12 months in treating patients who have stage III or stage IV ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of continuing paclitaxel for 12 months versus 3 months on progression free survival and overall survival in women with advanced ovarian, fallopian tube, or peritoneal cancer who attained complete remission on initial platinum (carboplatin or cisplatin) and paclitaxel based chemotherapy. II. Assess the toxic effects associated with prolonged paclitaxel administration in these patients.

OUTLINE: This is a randomized study. Patients are stratified by stage (optimal stage III vs suboptimal stage III vs stage IV), prior treatments with paclitaxel (over at least 24 hours vs over less than 24 hours), and age (65 and under vs over 65). Patients are randomized to one of two treatment arms. Arm I: Patients receive paclitaxel IV over 3 hours on day 1. Treatment continues every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive paclitaxel IV over 3 hours on day 1. Treatment continues every 4 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until disease progression or 1 year from registration, then every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 450 patients (225 per arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced ovarian epithelial, fallopian tube, or primary peritoneal cancer Must have undergone an initial exploratory laparotomy with tumor debulking AND Must be FIGO stage IIIA, IIIB, IIIC, or IV at the time of initial laparotomy Must have attained a clinically defined complete remission (CR) following treatment with platinum (cisplatin or carboplatin) and paclitaxel based combination chemotherapy regimen by achieving the following: No evidence of cancer on physical examination CA-125 no greater than 35 units/mL Creatinine no greater than 2.0 mg/dL OR Creatinine clearance greater than 60 mL/min Bilirubin no greater than 2.0 mg/dL Negative ascites No evidence of residual cancer on CT scan of the abdomen/pelvis or chest x-ray (or chest CT scan, if performed) No symptoms felt to be secondary to persistent malignancy Must have received a minimum of 5 and a maximum of 6 courses of chemotherapy prior to study Must register for study within 21 to 56 days after prior chemotherapy Not concurrently registered to SWOG-S9618, SWOG-S9619, SWOG-S9912, or SWOG-S0009 or front line treatment phase III GOG trials

PATIENT CHARACTERISTICS: Age: Any age Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,200/mm3 Platelet count at least 100,000/mm3 Hepatic: See Disease Characteristics Renal: See Disease Characteristics Other: No prior malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or incidental carcinoid

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent antitumor treatment No concurrent immunotherapy Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy Prior cisplatin allowed if initial dose at least 50 mg/m2 Prior carboplatin allowed if initial dose at least 300 mg/m2 or AUC at least 4 No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: No concurrent radiotherapy No prior abdominal/pelvic irradiation Surgery: See Disease Characteristics No second look laparotomy or laparoscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 1997-11; Primary Completion 2003-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
progression-free survival | duration between date of enrollment and date first recurrence or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Maurie Markman, MD, Study Chair — The Cleveland Clinic
Locations (93):
- United States (93):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Scripps Clinic Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Background] Markman M, Liu PY, Rothenberg ML, Monk BJ, Brady M, Alberts DS. Pretreatment CA-125 and risk of relapse in advanced ovarian cancer. J Clin Oncol. 2006 Mar 20;24(9):1454-8. doi: 10.1200/JCO.2005.04.7373. PMID 16549840
- [Background] Liu PY, Alberts DS, Monk BJ, et al.: Relationship between pretreatment CA-125 level and risk of relapse in advanced ovarian cancer (AOC) patients in a complete clinical response (CCR) who received "maintenance therapy". [Abstract] J Clin Oncol 23 (Suppl 16): A-5013, 458s, 2005.
- [Result] Liu PY, Alberts DS, Monk BJ, Brady M, Moon J, Markman M. An early signal of CA-125 progression for ovarian cancer patients receiving maintenance treatment after complete clinical response to primary therapy. J Clin Oncol. 2007 Aug 20;25(24):3615-20. doi: 10.1200/JCO.2006.09.4540. PMID 17704410
- [Result] Markman M, Liu P, Wilczynski S, et al.: Survival (S) of ovarian cancer (OC) patients (pts) treated on SWOG9701/GOG178: 12 versus (v) 3 cycles (C) of monthly single-agent paclitaxel (PAC) following attainment of a clinically-defined complete response (CR) to platinum (PLAT)/PAC. [Abstract] J Clin Oncol 24 (Suppl 18): A-5005, 257s, 2006.
- [Result] Markman M. Maintenance chemotherapy in advanced ovarian cancer: the US experience. Int J Gynecol Cancer. 2008 Mar-Apr;18 Suppl 1:40-3. doi: 10.1111/j.1525-1438.2007.01104.x. PMID 18336399
- [Result] Markman M, Liu PY, Wilczynski S, Monk B, Copeland LJ, Alvarez RD, Jiang C, Alberts D; Southwest Oncology Group; Gynecologic Oncology Group. Phase III randomized trial of 12 versus 3 months of maintenance paclitaxel in patients with advanced ovarian cancer after complete response to platinum and paclitaxel-based chemotherapy: a Southwest Oncology Group and Gynecologic Oncology Group trial. J Clin Oncol. 2003 Jul 1;21(13):2460-5. doi: 10.1200/JCO.2003.07.013. PMID 12829663